CLINICAL TRIAL: NCT01585870
Title: A Phase 1, Multi-center, Non-randomized, Open Label, Dose Escalation Design Study of Sorafenib (BAY43-9006) in Combination With Eribulin in Subjects With Advanced, Metastatic or Refractory Solid Tumors
Brief Title: Safety, Pharmacokinetics, Pharmacodynamics and Anti-tumor Activity of Sorafenib and Eribulin in Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Onyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15977; 2011-005849-12 (EudraCT Number)
Record Dates: First submitted 2012-04-12; First posted 2012-04-26 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Neoplasms
Keywords: Safety; Tolerability; Pharmacokinetics; Clinical benefit; Sorafenib; Eribulin; advanced metastatic solid tumors
MeSH Terms: conditions — Neoplasms | interventions — Sorafenib; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib + Eribulin (Experimental)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006); Drug: Eribulin

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib (starting dose of 200 mg bid, level 1) administration will begin on Day 11 of Cycle 1, and will be administered twice daily continuously. If the combination is well tolerated, the dose will be escalated in new cohorts to 200 mg AM and 400 mg PM (level 2), then subsequently to 400 mg bid (level 3).
  If sorafenib starting dose (level 1) is not well tolerated with eribulin, the sorafenib dose will be de-escalated to 200 mg qd (Dose Level -1) in a new cohort.
Drug: Eribulin — Eribulin: 1.4 mg/m2 as an intravenous infusion on Days 1 and 8 of each 21-day cycle.

SUMMARY:
This Phase 1 study will be conducted in an open-label, non-randomized, dose-escalation design in subjects with advanced, metastatic or refractory solid malignancy who are not candidates for standard therapy. The study drugs are sorafenib and eribulin mesylate.

Up to 24 subjects with solid tumors will participate in the dose escalation part of the study, and once the maximum tolerated dose is defined, up to 30 subjects with advanced, metastatic or refractory solid tumors will participate in the expansion phase of the study.

Eribulin (mesylate) will be administered intravenously at a fixed dose of 1.4 mg/m2 on Days 1 and 8 of 21-day Cycles.

The starting sorafenib dose (Dose Level 1) is 200 mg twice daily. Sorafenib is given orally, continuously on days 11 to 21 of Cycle 1, and from Day 1 to Day 21 of all subsequent cycles. If 200 mg sorafenib twice daily is tolerated with eribulin, the sorafenib dose will be escalated sequentially to 200 mg morning dose and 400 mg evening dose (Dose Level 2) in a new cohort. If Dose Level 2 is tolerated, a second dose escalation to 400 mg twice daily (Dose Level 3) will be studied in a new cohort. If the starting dose of sorafenib is not tolerated with eribulin, the sorafenib dose will be de-escalated to 200 mg once daily in a new cohort. Subjects will need to receive two cycles of eribulin plus sorafenib therapy and safety data for the first and second cycle needs to be available before the start of the next cohort.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced, metastatic or refractory solid malignancy who are not candidates for standard therapy. For subject with metastatic breast cancer, prior therapy should have included an anthracycline and a taxane in either the adjuvant or metastatic setting.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate bone marrow, cardiac, liver, renal and pancreatic function
* Predicted life expectancy of at least 12 weeks

Exclusion Criteria:

* Prolonged corrected QT (QTc), defined as QTcF (QT interval corrected for heart rate according to Fridericia) interval > 450 msec at screening by central reader
* Cardiac disease: Congestive heart failure > NYHA Class II; subjects must not have unstable angina (angina symptoms at rest) or new-onset angina (began within the last 3 months) or myocardial infarction within the past 6 months; cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Arterial or venous thrombi, including cerebrovascular accident and myocardial infarction in the past 6 months
* Pulmonary hemorrhage event ≥ CTCAE (common toxicity criteria for adverse events) Grade 2 within 4 weeks
* Any other hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks
* Chemotherapy, hormonal therapy, investigational drugs, or radiotherapy within the last 28 days and/or not recovered (< Grade 1) from prior therapy. Start of study treatment is allowed within less than 28 days of the prior therapy provided that 5 half-lives of the prior treatment drug(s) have elapsed.
* Use of medication that may prolong QTc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events as a Measure of Safety and Tolerability | Up to 30 months
AUC (area under the plasma concentration vs time curve) of BAY43-9006 | Up to 9 weeks
Cmax (maximum drug concentration in plasma after single dose administration) of BAY43-9006 | Up to 9 weeks
QT time, assessed by QTcF / QTcB (QT interval corrected for heart rate according to Fridericia / Bazett) | Up to 9 weeks

SECONDARY OUTCOMES:
Clinical benefit and response measured by RESIST (1.1) criteria | Approximately 3-18 weeks depending on tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Toulouse, France
- Germany (3):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Berlin, State of Berlin